CLINICAL TRIAL: NCT05863871
Title: Real World Study of Linperlisib for Lymphoma Treatment: Multicenter, Non-interventional and Observational Real-world Study
Brief Title: Real World Study of Linperlisib for Lymphoma Treatment
Acronym: MA-LYM-RWS-001
Status: Not yet recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Collaborators: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, M.D. and Ph.D, Ruijin Hospital
Other Study IDs: E20230190
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Focus on the Lymphoma Including B/T-cell Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- all enrolled patients: All patient who signed the consent form for participation to the study
  Interventions: Drug: Linperlisib

INTERVENTIONS:
Drug: Linperlisib — 80 mg, qd
  Other Names: YY-20394

SUMMARY:
This is a multicenter, non-interventional and observational real-world study to evaluate the efficacy and safety of linperlisib in patients with lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Clinical diagnosis of lymphoma patients
3. Patients signed informed consent, volunteered to join the study, and had the willingness and ability to cooperate with the data collection in this study;
4. The researchers' assessment can use Linperlisib treatment

Exclusion Criteria:

1. The nature of the study could not be understood or informed consent was not obtained
2. Other ineligible conditions were assessed by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical diagnosis of lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse events (AEs)/ serious adverse events (SAEs) | up to 4 weeks after the last dose
  Rate of adverse events (AEs)/ serious adverse events (SAEs) in patients with lymphoma receiving linperlisib therapy

SECONDARY OUTCOMES:
Complete response rate | 6 months
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Progression-free survival | 1 years and 2 years
  Progression-free survival was defined as the time from the date of enrollment until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Overall survival | Baseline up to data cut-off (up to approximately 2 years)
  Overall survival was defined as the time from the date of enrollment to the date of death from any cause.
Duration of response | Baseline up to data cut-off (up to approximately 2 years)
  Duration of response was defined as the time from the date of favorable response until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Tianjin Cancer Hospital/ Tianjin medical university cancer institute & hospital, Tianjin

IPD SHARING:
Plan to Share IPD: Undecided
The safty of Linperlisib in lymphoma patients